CLINICAL TRIAL: NCT00133237
Title: Prospective, Randomized Trial of the Sirolimus-Eluting Stent and Paclitaxel-Eluting Stent for the Treatment of Unprotected Left Main Coronary Artery Disease(ISAR-LEFT-MAIN)
Brief Title: Drug-eluting-stents for Unprotected Left Main Stem Disease (ISAR-LEFT-MAIN)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Collaborators: Technical University of Munich (Other)
Responsible Party: Albert Schömig, Deutsches Herzzentrum Muenchen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE No. S02005
Record Dates: First submitted 2005-08-22; First posted 2005-08-23 (Estimated); Last update posted 2010-03-15 (Estimated); Status verified 2008-10

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Sirolimus-eluting stent (Cypher)
  Interventions: Device: Sirolimus-eluting stent
- B (Active Comparator): Paclitaxel-eluting stent (Taxus)
  Interventions: Device: Paclitaxel-eluting stent

INTERVENTIONS:
Device: Sirolimus-eluting stent — cypher stent is implanted due to randomization.
  Other Names: Cypher
  Arms: A
Device: Paclitaxel-eluting stent — taxus stent is implanted due to randomization.
  Other Names: Taxus
  Arms: B

SUMMARY:
The purpose of this study is to evaluate the efficacy of sirolimus- and paclitaxel-eluting stents for treatment of unprotected left main coronary artery disease.

DETAILED DESCRIPTION:
With the advent of coronary stents and improvements in periprocedural antithrombotic regimen, the spectrum of indications of percutaneous coronary interventions has continuously expanded for patients with coronary heart disease, gaining ground in what have been traditionally considered as domains of coronary bypass surgery. Several groups reported the outcomes of patients with unprotected left main coronary artery (LMCA) disease treated with stenting. Most of them found that LMCA stenting was feasible and safe, and, in low-risk patients, it was associated with minimal periprocedural complications and low long-term morbidity and mortality. Despite these encouraging reports, a widespread use of this technique has been hampered by the still high incidence of restenosis. It is commonly accepted that coronary bypass graft surgery and stenting for unprotected LMCA disease are associated with similar rates of mortality, and that the higher incidence of restenosis and greater need for revascularization procedures after LMCA stenting remain the major contributors for the observed difference in clinical efficacy between both therapies. The recent introduction of stents eluting anti-restenotic drugs, with sirolimus and paclitaxel the most studied compounds, has opened new perspectives for the prevention of restenosis. Several randomized trials have reported excellent results in the reduction of restenosis and need for reinterventions with drug-eluting stents (DES). Although, none of these trials studied the benefit of DES for lesions located in the LMCA, their results suggested that use of these new devices may be particularly helpful for the reduction of restenosis in the group of patients with left main trunk disease. This is supported by the findings of several series of patients with unprotected LMCA disease who have been successfully treated with DES. Importantly, for patients who are unable to undergo CABG due to cardiac surgeons' refusal (poor surgical candidates) or their own unwillingness, stenting with DES remains the only revascularization alternative. Recent guidelines of PCI recommend stenting, preferentially with DES, for unprotected LMCA in the absence of other revascularization options.

Comparison:

Sirolimus-eluting stents compared with paclitaxel-eluting stent for treatment of lesions allocated at left main trunk.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than age 18 with ischemic symptoms or evidence of myocardial ischemia in the presence of ≥50% stenosis located in unprotected LMCA who are unable to undergo coronary artery bypass graft (CABG)
* Pretreatment with a loading dose of 300-600 mg clopidogrel
* Informed, written consent

Exclusion Criteria:

* Cardiogenic shock;
* ST-segment elevation acute myocardial infarction within 48 h from symptom onset;
* In-stent restenosis;
* Malignancies or other comorbid conditions with life expectancy less than one year;
* Prior coronary artery bypass surgery with revascularization of left anterior descending (LAD) and/or left circumflex (LCx) coronary artery
* Planned staged percutaneous coronary intervention (PCI) procedure within 30 days from index procedure or prior PCI within the last 30 days
* Left main size >4.5mm
* An elective surgical procedure is planned during the first six months post enrolment;
* Known allergy to the study medications
* Pregnancy
* Patient's inability to fully cooperate with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 607 (Actual)
Dates: Start 2005-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac events (composite of death, myocardial infarction and target lesion revascularization) at one year | one year

SECONDARY OUTCOMES:
Angiographic restenosis at 6-9 month follow-up angiography (based on left main area analysis) | 6-9 months

CONTACTS AND LOCATIONS:
Overall Officials: Albert Schömig, MD, Study Chair — Deutsches Herzzentrum Muenchen; Adnan Kastrati, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (2):
- Germany (2):
  - Deutsches Herzzentrum, Munich
  - First Medizinische Klinik, Klinikum rechts der Isar, Munich

REFERENCES:
- [Background] Ellis SG, Tamai H, Nobuyoshi M, Kosuga K, Colombo A, Holmes DR, Macaya C, Grines CL, Whitlow PL, White HJ, Moses J, Teirstein PS, Serruys PW, Bittl JA, Mooney MR, Shimshak TM, Block PC, Erbel R. Contemporary percutaneous treatment of unprotected left main coronary stenoses: initial results from a multicenter registry analysis 1994-1996. Circulation. 1997 Dec 2;96(11):3867-72. doi: 10.1161/01.cir.96.11.3867. PMID 9403609
- [Background] Park SJ, Park SW, Hong MK, Cheong SS, Lee CW, Kim JJ, Hong MK, Mintz GS, Leon MB. Stenting of unprotected left main coronary artery stenoses: immediate and late outcomes. J Am Coll Cardiol. 1998 Jan;31(1):37-42. doi: 10.1016/s0735-1097(97)00425-7. PMID 9426015
- [Background] Takagi T, Stankovic G, Finci L, Toutouzas K, Chieffo A, Spanos V, Liistro F, Briguori C, Corvaja N, Albero R, Sivieri G, Paloschi R, Di Mario C, Colombo A. Results and long-term predictors of adverse clinical events after elective percutaneous interventions on unprotected left main coronary artery. Circulation. 2002 Aug 6;106(6):698-702. doi: 10.1161/01.cir.0000024983.34728.5d. PMID 12163430
- [Background] Ellis SG, Hill CM, Lytle BW. Spectrum of surgical risk for left main coronary stenoses: benchmark for potentially competing percutaneous therapies. Am Heart J. 1998 Feb;135(2 Pt 1):335-8. doi: 10.1016/s0002-8703(98)70102-4. PMID 9489985
- [Background] Chieffo A, Stankovic G, Bonizzoni E, Tsagalou E, Iakovou I, Montorfano M, Airoldi F, Michev I, Sangiorgi MG, Carlino M, Vitrella G, Colombo A. Early and mid-term results of drug-eluting stent implantation in unprotected left main. Circulation. 2005 Feb 15;111(6):791-5. doi: 10.1161/01.CIR.0000155256.88940.F8. Epub 2005 Feb 7. PMID 15699254
- [Background] Valgimigli M, van Mieghem CA, Ong AT, Aoki J, Granillo GA, McFadden EP, Kappetein AP, de Feyter PJ, Smits PC, Regar E, Van der Giessen WJ, Sianos G, de Jaegere P, Van Domburg RT, Serruys PW. Short- and long-term clinical outcome after drug-eluting stent implantation for the percutaneous treatment of left main coronary artery disease: insights from the Rapamycin-Eluting and Taxus Stent Evaluated At Rotterdam Cardiology Hospital registries (RESEARCH and T-SEARCH). Circulation. 2005 Mar 22;111(11):1383-9. doi: 10.1161/01.CIR.0000158486.20865.8B. PMID 15781749
- [Background] Silber S, Albertsson P, Aviles FF, Camici PG, Colombo A, Hamm C, Jorgensen E, Marco J, Nordrehaug JE, Ruzyllo W, Urban P, Stone GW, Wijns W; Task Force for Percutaneous Coronary Interventions of the European Society of Cardiology. Guidelines for percutaneous coronary interventions. The Task Force for Percutaneous Coronary Interventions of the European Society of Cardiology. Eur Heart J. 2005 Apr;26(8):804-47. doi: 10.1093/eurheartj/ehi138. Epub 2005 Mar 15. PMID 15769784
- [Result] Mehilli J, Kastrati A, Byrne RA, Bruskina O, Iijima R, Schulz S, Pache J, Seyfarth M, Massberg S, Laugwitz KL, Dirschinger J, Schomig A; LEFT-MAIN Intracoronary Stenting and Angiographic Results: Drug-Eluting Stents for Unprotected Coronary Left Main Lesions Study Investigators. Paclitaxel- versus sirolimus-eluting stents for unprotected left main coronary artery disease. J Am Coll Cardiol. 2009 May 12;53(19):1760-8. doi: 10.1016/j.jacc.2009.01.035. PMID 19422982
- [Derived] Cassese S, Kufner S, Xhepa E, Byrne RA, Kreutzer J, Ibrahim T, Tiroch K, Valgimigli M, Tolg R, Fusaro M, Schunkert H, Laugwitz KL, Mehilli J, Kastrati A. Three-year efficacy and safety of new- versus early-generation drug-eluting stents for unprotected left main coronary artery disease insights from the ISAR-LEFT MAIN and ISAR-LEFT MAIN 2 trials. Clin Res Cardiol. 2016 Jul;105(7):575-84. doi: 10.1007/s00392-015-0953-x. Epub 2015 Dec 22. PMID 26689707
- [Derived] Tiroch K, Mehilli J, Byrne RA, Schulz S, Massberg S, Laugwitz KL, Vorpahl M, Seyfarth M, Kastrati A; ISAR-LEFT MAIN Study Investigators. Impact of coronary anatomy and stenting technique on long-term outcome after drug-eluting stent implantation for unprotected left main coronary artery disease. JACC Cardiovasc Interv. 2014 Jan;7(1):29-36. doi: 10.1016/j.jcin.2013.08.013. Epub 2013 Dec 11. PMID 24332416